CLINICAL TRIAL: NCT00724009
Title: Clofarabine Bone Marrow Cytoreduction : Feasibility of Induction as a Bridge to Allogeneic Stem Cell Transplantation for Patients With Relapsed or Refractory Acute Leukemias, Myelodysplastic Syndromes, and Advanced Myeloproliferative Diseases.
Brief Title: Clofarabine Bone Marrow Cytoreduction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15809B
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Results first posted 2014-03-18 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-01

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia | interventions — Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Clofarabine (Experimental): Clofarabine 30 mg/m2/day IV infusion over one hour for 5 consecutive days
  Interventions: Drug: Clofarabine

INTERVENTIONS:
Drug: Clofarabine — Clofarabine for injection should be diluted with 0.9% sodium chloride injection USP or European Pharmacopeia (EP) normal saline (NS) or 5% dextrose injection (D5W) USP or EP prior to IV infusion. The resulting admixture may be stored at room temperature, but must be used within 24 hours of preparation. Clofarabine should be diluted with NS or D5W prior to administering by IV infusion. The dosage is based on the patient's body surface area (BSA), calculated using the actual height and weight before the start of each cycle. To prevent drug incompatibilities, no other medications should be administered through the same IV line.
  Other Names: Clolar

SUMMARY:
For relapsed and refractory leukemia patients induction chemotherapy prior to initiating a conditioning regimen will decrease residual leukemia (as measured by bone marrow leukemia blast percentage) at the time of HCT. This should lead to reduced relapse while still maintaining low transplant related mortality.

DETAILED DESCRIPTION:
Screening will be done prior to enrollment in the study. The following will be done as part of the screening process:

* Medical history review
* Physical exam
* Measurement of vital Signs
* Blood tests (approximately 6 teaspoons of blood) will be done to see if the liver and kidneys are healthy, HIV (the virus that causes AIDS) test for this study and pregnancy test.
* Urine test
* Bone marrow biopsy and aspirate

If the patient is ineligible or does not have a donor for Allogeneic Stem Cell transplantation, you will not be able to participate in this clinical trial.

After results of these tests are obtained, your doctor will decide whether you can participate in this study.

Study procedures:

The study drug will be given for 5 days.

Days 1 through 5:

The patient will receive dexamethasone 1.5 hours prior to the administration of Clofarabine as part of standard care for subjects receiving Clofarabine.

The patient will receive an intravenous (IV) injection (into the vein) of Clofarabine each day for 5 days. This injection is given in the hospital and will be given over approximately 60 minutes each day. The actual dose of Clofarabine is based on the weight and height of the subject.

The patient will have the following tests done to see the effects of the study drug:

Each day of Clofarabine administration, on day 12 and then each day until stem cell transplantation:

* Physical exam
* Vital signs
* Blood tests. About 3-4 teaspoons will be taken each time.

Day 12 after Clofarabine administration and then as outlined for stem cell transplantation:

• Bone marrow biopsy and aspirate.

After Clofarabine administration, there will be short resting period of 7-14 days. After the resting period, the patient will start receiving conditioning chemotherapy regimen (other standard of care drugs to better prepare your body for the stem cell transplant). This regimen will begin 15-21 days after they first received Clofarabine, and consists of additional treatment (chemotherapy and/or radiation). The type of treatment(s) the patient will receive for conditioning is dependent on the type of disease. In addition, this treatment will be decided by your doctor and is independent of this research. The duration of the conditioning period is variable and may take between 5-8 days. Stem cells are usually given one day after the completion of this regimen, which will be between 21 and 30 days after the patient has first received Clofarabine.

Follow-up Subjects who have a response and proceed with stem cell transplant will be followed weekly for the first three months and then every month for six months, then every two months for 12 months, then every three months for 18 months. The stem cell transplant will be done 21-30 days after first receiving Clofarabine. Subjects who do not go on to stem cell transplant will be followed for 3 months following administration of Clofarabine.

At these visits, the following will be done:

* A physical exam
* Medical history
* Blood tests (about 3 teaspoons blood will be taken) performed.

End of study

At this time, the following tests will be done:

* Physical exam
* Blood tests
* Bone marrow biopsy

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent.
* Adequate hepatobiliary function as indicated by the following laboratory values:

  * SGOT/SGPT <=2.5 x upper limit of normal
  * Alkaline phosphatase <=2.5 x upper limit of normal
  * Serum bilirubin < 1.5 mg/dl
  * Adequate renal function as indicated by the following laboratory values:
  * Creatinine Clearance >50 ml/min
* Age >/=18 years
* Zebroid performance status </= 2 (See Appendix A)
* Life expectancy is not severely limited by concomitant illness (i.e. < 3months life expectancy from non-leukemic conditions).
* No evidence of chronic active hepatitis or cirrhosis.
* HIV-negative
* Male and female patients must use an effective contraceptive method during the study and for a minimum of 6 months after study treatment.
* Female patients of childbearing potential must have a negative serum pregnancy test within 2 weeks prior to enrollment.

Exclusion Criteria:

* Current concomitant chemotherapy, radiation therapy, or immunotherapy other than as specified in the protocol.
* Use of investigational agents within 30 days or any anticancer therapy within 2 weeks before study entry with the exception of hydroxyurea. The patient must have recovered from all acute non-hematologic toxicities from any previous .
* Have any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver, or other organ system that may place the patient at undue risk to undergo treatment.
* Patients with a systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
* Pregnant or lactating patients.
* Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-12; Primary Completion 2010-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Stock, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago hospitals, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clofarabine
Started | 29
Completed | 29 (One patient underwent conditioning but died 1 day before stem cell infusion due to sepsis.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Clofarabine
Number analyzed (Participants) | 29
Age, Continuous [Median (Full Range); unit: years] | 51 [23 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Cytoreductive Response
Description: Percent of patients achieving cytoreductive response of marrow cellularity <20% and blasts < 10%
Time Frame: Day 12
Measure: Number; unit: percentage of participants
Arm/Group | Clofarabine
Number analyzed (Participants) | 29
percentage of participants | 52

2. Secondary Outcome: Number of Participants With Renal Adverse Events
Description: Treatment-related toxicity was calculated according to Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.
Time Frame: Day 12
Measure: Number; unit: participants
Arm/Group | Clofarabine
Number analyzed (Participants) | 29
participants
  Grade 1-2 | 9
  Grade 3-4 | 1

3. Secondary Outcome: Number of Participants With Hepatic (Total Bilirubin) Adverse Events
Description: as for outcome 2
Time Frame: Day 12
Measure: Number; unit: participants
Arm/Group | Clofarabine
Number analyzed (Participants) | 29
participants
  Grade 1-2 | 14
  Grade 3-4 | 3

4. Secondary Outcome: Number of Participants With Hepatic (SGOT) Adverse Events
Description: as for outcome 2
Time Frame: Day 12
Measure: Number; unit: participants
Arm/Group | Clofarabine
Number analyzed (Participants) | 29
participants
  Grade 1-2 | 14
  Grade 3-4 | 9

5. Secondary Outcome: Number of Participants With Cardiac Adverse Events
Description: as for outcome 2
Time Frame: Day 12
Measure: Number; unit: participants
Arm/Group | Clofarabine
Number analyzed (Participants) | 29
participants
  Grade 1-2 | 2
  Grade 3-4 | 0

6. Secondary Outcome: Number of Participants With Skin Adverse Events
Description: as for outcome 2
Time Frame: Day 12
Measure: Number; unit: participants
Arm/Group | Clofarabine
Number analyzed (Participants) | 29
participants
  Grade 1-2 | 1
  Grade 3-4 | 0

7. Secondary Outcome: Number of Participants Infection Adverse Events
Description: as for outcome 2
Time Frame: Day 12
Measure: Number; unit: participants
Arm/Group | Clofarabine
Number analyzed (Participants) | 29
participants
  Grade 3-4 | 11
  Grade 5 | 1

8. Secondary Outcome: Leukemia Free Survival
Description: Time to event analysis used the day of transplant as day 0.
Time Frame: 2 years
Population: One patient with refractory AML underwent conditioning but died 1 day before stem cell infusion due to sepsis (grade 5 infection)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Clofarabine
Number analyzed (Participants) | 28
days | 211 [171 to 342]

ADVERSE EVENTS:
Arm/Group | Clofarabine
Serious Adverse Events (participants affected / at risk) | 22/29
Other Adverse Events (participants affected / at risk) | 26/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clofarabine (N=29)
Renal (creatine) (Renal and urinary disorders) | 1 (1)
Hepatic (total bilirubin) (Hepatobiliary disorders) | 3 (3)
Hepatic (SGOT) (Hepatobiliary disorders) | 9 (9)
Infection (Infections and infestations) | 12 (12)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clofarabine (N=29)
Renal (creatinine) (Renal and urinary disorders) | 9 (9)
Hepatic (total bilirubin) (Hepatobiliary disorders) | 14 (14)
Hepatic (SGOT) (Hepatobiliary disorders) | 14 (14)
Cardiac (Cardiac disorders) | 2 (2)
Skin (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No